CLINICAL TRIAL: NCT04507399
Title: Investigating Consumers Perception and Acceptance of Whey Beverages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Lisa Methven, Head of Sensory Science, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: SCFP 32/20
Record Dates: First submitted 2020-07-25; First posted 2020-08-11 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Individual Difference; Food Sensitivity; Food Preferences
Keywords: Mouthdrying; Saliva Flow; Mucoadhesion; Oral Nutritional Supplements
MeSH Terms: conditions — Food Intolerance; Food Preferences

STUDY DESIGN:
Intervention Model Description: This study involves both a crossover design where each participant tastes both the control product and the protein fortified product with an appropriate break between the two sessions. The study will be conducted single blind as it not feasible to blind the researcher. Each participant will attend 2 study visits and all foods will be presented with random blinding codes.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein Beverage (Experimental): Whey Protein Beverage
  Interventions: Behavioral: Liquid Model
- Control Beverage (Experimental): Whey Permeate Beverage
  Interventions: Behavioral: Liquid Model

INTERVENTIONS:
Behavioral: Liquid Model — To study the perception of whey beverages using sensory methods (rating drying as well as discrimination tests "which is the stronger in drying")
  Measuring mucoadhesion via protein content remaining in saliva following swallowing of whey protein and whey permeate beverages.

SUMMARY:
Brief Summary: This study aims to investigate whether protein fortification of beverages causes mouthdrying and mucoadhesion and whether this is influenced by saliva flow.

DETAILED DESCRIPTION:
To investigate whether whey protein beverages causes mouthdrying and reduces acceptability compared with a control beverage (whey permeate beverage) and to determine whether manipulating salivary flow rates influences mouthdrying.

To determine whether mucoadhesion is a probable cause of mouthdrying.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* No food allergies or intolerances
* Non smokers

Exclusion Criteria:

* Taking prescribed medication that could influence study outcomes (such as saliva flow)
* Relevant food allergies or intolerances
* Outside age criteria
* Cancer
* Had oral surgery or a stroke
* Smoker
* Diabetic
* Anyone who currently has COVID-19 symptoms or who has had COVID-19 within the last 4 weeks

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Mucoadhesion and Mouthdrying | Saliva collection and mouthdrying scoring throughout visits, 2 days
  Following swallowing of different whey beverage samples (whey protein / whey permeate), volunteers will be asked either to rate samples for mouthdrying or to spit their saliva into a tube at specific timepoints (15s & 60s) with appropriate rest periods. The rating and spitting times will be set within a balanced order protocol.

SECONDARY OUTCOMES:
Mouthdrying from whey beverages | 1 day (Sampled at study visit one)
  Perceived mouth drying from whey beverages (whey permeate / whey protein) using data from sensory methods (rating drying as well as discrimination tests "which is the stronger in drying"). Scale for scoring is the gLMS scale (general linear magnitude scale); higher value is worse outcome.
Manipulating saliva flow and mouthdrying from whey beverages | 1 day (Sampled at study visit one)
  Volunteers will be asked to manipulate their saliva flow and consume whey beverages (whey permeate / whey protein) and score perceived mouth drying (data will be collected from sensory methods (rating drying as well as discrimination tests "which is the stronger in drying")
Saliva collection | 1 day (Sampled at study visit two)
  Salivary flow rates from unstimulated and stimulated saliva samples.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Methven, Principal Investigator — University of Reading
Locations (1):
- Sensory Science Centre, Department of Food and Nutritional Science, University of Reading, Reading, Berkshire, United Kingdom, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however it is possible that some of the individual (unliked / non identifiable) data will be useful in a meta analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Bull SP, Hong Y, Khutoryanskiy VV, Parker JK, Faka M, Methven L. Whey protein mouth drying influenced by thermal denaturation. Food Qual Prefer. 2017 Mar;56(Pt B):233-240. doi: 10.1016/j.foodqual.2016.03.008. PMID 28260840
- [Background] Withers CA, Cook MT, Methven L, Gosney MA, Khutoryanskiy VV. Investigation of milk proteins binding to the oral mucosa. Food Funct. 2013 Nov;4(11):1668-74. doi: 10.1039/c3fo60291e. PMID 24092277
- [Background] Affoo RH, Foley N, Garrick R, Siqueira WL, Martin RE. Meta-Analysis of Salivary Flow Rates in Young and Older Adults. J Am Geriatr Soc. 2015 Oct;63(10):2142-51. doi: 10.1111/jgs.13652. Epub 2015 Oct 12. PMID 26456531
- [Background] Withers CA, Lewis MJ, Gosney MA, Methven L. Potential sources of mouth drying in beverages fortified with dairy proteins: A comparison of casein- and whey-rich ingredients. J Dairy Sci. 2014 Mar;97(3):1233-47. doi: 10.3168/jds.2013-7273. Epub 2014 Jan 17. PMID 24440265